CLINICAL TRIAL: NCT07309432
Title: A Randomized, Double-Masked, Placebo-Controlled, Phase 3 Study to Assess the Efficacy and Safety of Bet v 1 Monoclonal Antibodies in Participants With Allergic Conjunctivitis Due to Birch Pollen Allergy
Brief Title: Study of Bet v1 Antibodies Effect on Eye Allergy Symptoms in Adolescents and Adults With Birch Pollen Allergy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5713-5715-ALG-2556
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Allergic Conjunctivitis
Keywords: Birch Pollen Allergy; Ocular allergy symptoms; Ocular allergy signs
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- REGN5713-5715 (Experimental)
  Interventions: Drug: REGN5713; Drug: REGN5715
- REGN5713 (Experimental)
  Interventions: Drug: REGN5713
- REGN5715 (Experimental)
  Interventions: Drug: REGN5715
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN5713 — Administered per protocol
  Other Names: Bremzalerbart
  Arms: REGN5713; REGN5713-5715
Drug: REGN5715 — Administered per protocol
  Other Names: Atisnolerbart
  Arms: REGN5713-5715; REGN5715
Drug: Placebo — Administered per protocol
  Arms: Placebo

SUMMARY:
This study is researching 2 experimental drugs, REGN5713 and REGN5715. The study drugs will be either of these drugs given alone (either REGN5713 or REGN5715) or given together (REGN5713 and REGN5715) to reduce eye allergy signs and symptoms due to birch tree pollen allergy.

The aim of the study is to see how safe and effective the study drugs are at lowering eye allergy signs and symptoms compared with placebo.

The study will also evaluate whether the combination (REGN5713-5715) has different effectiveness than REGN5713 or REGN5715 alone.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* How much of the study drugs is in the blood at different times
* Whether the body makes antibodies against the study drugs (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Positive SPT to birch allergen extract
2. Positive allergen specific Immunoglobulin E (sIgE) tests for birch and Bet v 1
3. Positive CAC criteria

Key Exclusion Criteria:

1. Significant and/or severe environmental allergies causing symptoms (outside of the challenge setting) that are expected to interfere with study assessments
2. Presence of any ophthalmic disease/abnormality/condition that may interfere with study assessments, affect the study outcomes or negatively impact participant safety
3. A clinical history of asthma with treatment of asthma requiring systemic (oral or parenteral) corticosteroid treatment more than twice within prior 12 months or once within 3 months prior to screening visit 1 or has been hospitalized or has attended the Emergency Room/Urgent Care facility for asthma in the 12 months prior to screening

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Ocular itch score in participants receiving REGN5713-5715 compared to placebo | At Day 8 post-Conjunctival Allergen Challenge (CAC)
  Assessed using the Ora Calibra® Conjunctival Allergen Challenge Ocular Itching Scale, a 0-4 scale where 0 = none and 4= incapacitating itch, 0.5 unit increments

SECONDARY OUTCOMES:
Achievement of at least a 1-point reduction in ocular itch score for at least 2 out of 3 post-CAC time points in participants receiving REGN5713-5715 compared to placebo | Baseline to Day 8 post-CAC
Ocular itch score in participants receiving REGN5713-5715 compared to placebo | At Day 57 post-CAC
Conjunctival redness score in participants receiving REGN5713-5715 compared to placebo | At Day 8 and Day 57 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale] ciliary [ciliary redness scale], episcleral [episcleral redness scale] vessel beds), a 0 to 4 scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Achievement of at least a 1-point reduction in conjunctival redness score for at least 2 out of 3 post-CAC time points in participants receiving REGN5713-5715 compared to placebo | Baseline to Day 8 post-CAC
Total Nasal Symptom Score (TNSS) in participants receiving REGN5713-5715 compared to placebo | At Day 8 post-CAC
  The TNSS ranges from 0 to 12 and is based on assessment of 4 nasal symptoms graded on a verbal rating scale ranging from 0 (none) to 3 (severe) for nasal congestion, nasal itching, rhinorrhea, and sneezing.
Ocular itch score in participants receiving REGN5715 compared to placebo | At Day 8 and Day 57 post-CAC
Achievement of at least a 1-point reduction in ocular itch score for at least 2 out of 3 post-CAC time points in participants receiving REGN5715 compared to placebo | Baseline to Day 8 post-CAC
Conjunctival redness score in participants receiving REGN5715 compared to placebo | At Day 8 post-CAC
Achievement of at least a 1-point reduction in conjunctival redness score in for at least 2 out of 3 post-CAC time points participants receiving REGN5715 compared to placebo | Baseline to Day 8 post-CAC
Ocular itch score in participants receiving REGN5713 compared to placebo | At Day 8 and Day 57 post-CAC
Achievement of at least a 1-point reduction in ocular itch score for at least 2 out of 3 post-CAC time points in participants receiving REGN5713 compared to placebo | Baseline to Day 8 post-CAC
Conjunctival redness score in participants receiving REGN5713 compared to placebo | At Day 8 post-CAC
Achievement of at least a 1-point reduction in conjunctival redness score for at least 2 out of 3 post-CAC time points in participants receiving REGN5713 compared to placebo | Baseline to Day 8 post-CAC
Percent change in birch titrated Skin Prick Test (tSPT) in participants receiving REGN5713-5715 compared to placebo | Baseline and at Day 8 post-CAC
  Area Under the Curve (AUC) of the mean wheal diameters
Ocular itch score in participants receiving REGN5713-5715 compared to REGN5713 | Baseline to Day 8 post-CAC
Ocular itch score in participants receiving REGN5713-5715 compared to REGN5715 | Baseline to Day 8 post-CAC
Achievements of different response thresholds for the ocular itch score among participants receiving REGN5713-5715, REGN5713, REGN5715 or placebo | Baseline to Day 8 post-CAC
Achievement of at least a 1-point reduction in ocular itch score for at least 2 out of 3 post-CAC time points in participants receiving REGN5713-5715 compared to placebo | Baseline to Day 57 post-CAC
Achievement of at least a 1-point reduction in conjunctival redness score for at least 2 out of 3 post-CAC time points in participants receiving REGN5713-5715 compared to placebo | Baseline to Day 57 post-CAC
Ciliary redness score in participants receiving REGN5713-5715 compared to placebo | At Day 8 and Day 57 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale] ciliary [ciliary redness scale], episcleral [episcleral redness scale] vessel beds), a 0 to 4 scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Episcleral redness score in participants receiving REGN5713-5715 compared to placebo | At Day 8 and Day 57 post-CAC
  Assessed using the Ora Calibra® Hyperemia Scale (for conjunctival [conjunctival redness scale] ciliary [ciliary redness scale], episcleral [episcleral redness scale] vessel beds), a 0 to 4 scale, where 0 = none and 4 = extremely severe, 0.5 unit increments
Total redness score in participants receiving REGN5713-5715 compared to placebo | At Day 8 and Day 57 post-CAC
  The total redness score is calculated for CAC: range 0 to 12, where higher scores indicate worse responses (calculated as a sum of the bilateral averages for conjunctival redness score, graded 0 = none to 4 = extremely severe + ciliary redness score, graded 0 = none and 4 = extremely severe + episcleral redness score, graded 0 = none and 4 = extremely severe)
Percent change in birch tSPT in participants receiving REGN5713-5715 compared to placebo | Baseline and at Day 57 post-CAC
Percent change in birch tSPT in participants receiving REGN5715 compared to placebo | Baseline, at Day 8 and at Day 57 post-CAC
Percent change in birch tSPT in participants receiving REGN5713 compared to placebo | Baseline, at Day 8 and at Day 57 post-CAC
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Up to Day 113
Severity of TEAEs | Up to Day 113
Occurrence of Treatment Emergent-Serious Adverse Events (TE-SAEs) | Up to Day 113
Concentrations of total REGN5713 is serum over time | Up to Day 113
Concentrations of total REGN5715 is serum over time | Up to Day 113
Occurrence of Anti-Drug Antibodies (ADA) responses to REGN5713 | Up to Day 113
Magnitude of ADA to REGN5713 | Up to Day 113
Occurrence of ADA responses to REGN5715 | Up to Day 113
Magnitude of ADA to REGN5715 | Up to Day 113

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/